CLINICAL TRIAL: NCT07239323
Title: Intracellularly Prepared Chimeric Antigen Receptor T-cell Therapy Targeting CD19 for the Treatment of Relapsed/Refractory Hematological Malignancies
Brief Title: In VIVO CAR-T Therapy for Relapsed/Refractory Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC027-1
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: B-Acute Lymphoblastic Leukemia; B Cell Non-Hodgkin's Lymphoma; Multiple Myeloma
Keywords: in Vivo; CAR-T; malignant hematological tumors
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Invivo CAR-T (Experimental)
  Interventions: Biological: Invivo CAR-T

INTERVENTIONS:
Biological: Invivo CAR-T — Patients were enrolled and given a single dose of CAR-T injection intravenously, hospitalized for observation over the following month, and followed up for observation over the following 2 years.

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with relapsed or refractory malignant hematological tumors.

It is an early exploratory clinical study of the safety, tolerability and initial efficacy in the treatment of relapsed or refractory malignant hematological tumors.

DETAILED DESCRIPTION:
This is an open-label, single-arm study to evaluate the efficacy and safety of in vivo Chimeric Antigen Receptor T-Cell(CAR-T cell) therapy in patients with relapsed refractory malignant hematological tumors. Upon enrollment, subjects will receive an intravenous infusion of the in Vivo CAR-T preparation. Following the infusion, subjects will be hospitalized for observation, and subjects will be evaluated for safety and efficacy. Subjects will be followed for up to 2 years to determine if the disease is under control.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender unrestricted;
2. Confirmed diagnosis of relapsed/refractory malignant hematological tumors, including B-ALL, B-cell lymphoma and multiple myeloma;
3. ECOG performance status score 0-2, with an expected survival period of ≥ 3 months;
4. Blood routine test results during the screening period meet the following criteria:

   ① Hemoglobin ≥ 6 g/dL (no red blood cell transfusion within 1 week before screening), recombinant human erythropoietin (rhEPO) is allowed; for patients meeting the hemoglobin ≥ 6 g/dL criterion, red blood cell transfusion can be used to maintain hemoglobin ≥ 6 g/dL;
   * Absolute neutrophil count (ANC) ≥ 600/μL (no use of granulocyte colony-stimulating factor [G-CSF] within 1 week before screening, or no use of pegylated G-CSF within 2 weeks before screening); ③ Platelet count ≥ 50,000/μL; ④ Lymphocyte count ≥ 500/μL;
5. Normal renal function during the screening period: creatinine clearance rate (CrCl) ≥ 45 mL/min (calculated using the Cockcroft-Gault formula);
6. Liver function during the screening period meets the following criteria:

   ① Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3.0 × ULN;

   ② Total bilirubin (TBIL) ≤ 2.0 × ULN (except for congenital hyperbilirubinemia such as Gilbert's syndrome, direct bilirubin can be relaxed to ≤ 1.5 × ULN);
7. Cardiac function during the screening period meets the following criteria:

   ① Left ventricular ejection fraction (LVEF) ≥ 40% (measured by echocardiography or MUGA scan);

   ② No clinically significant pericardial effusion;

   ③ No clinically significant electrocardiogram (ECG) abnormalities;
8. Pulmonary function during the screening period meets the following criteria: blood oxygen saturation (SpO₂) ≥ 90%;
9. Women of childbearing age must have a negative pregnancy test during the screening period and before drug administration, and must not be in the lactation period;
10. Men and women of childbearing age must agree to take effective contraceptive measures and not donate reproductive cells (including sperm or eggs) from the time of signing the informed consent form until 1 year after the end of study drug administration;
11. The subject or their legally authorized representative has signed the informed consent form (ICF), indicating their understanding of the purpose and procedures of the study and their voluntary participation in this study.

Exclusion Criteria:

1. Other anti-tumor treatments within the screening period (judged by the investigator comprehensively):

   ① Received chemotherapy, targeted therapy or immunotherapy within 5 half-lives before administration;

   ② Received radiotherapy within 4 weeks before administration (if the radiotherapy target area covers ≤ 5% of bone marrow reserve, the time limit for radiotherapy completion is not restricted);
2. History of hematopoietic stem cell transplantation: Received allogeneic or autologous hematopoietic stem cell transplantation within 3 months before administration;
3. History of other malignant tumors (except for this disease), except for the following situations:

   ① Received radical treatment and had no known active disease for ≥ 2 years before enrollment;

   ② Had fully treated non-melanoma skin cancer in the past and had no active lesions at present;
4. Received treatment related to vesicular stomatitis virus glycoprotein (VSVG) pseudotyped virus in the past;
5. Had severe and uncontrolled infections (bacterial, viral, fungal, etc.) within the screening period;
6. Clinically significant cardiac diseases:

   * Had symptomatic heart failure or other serious cardiac diseases (such as severe arrhythmia);

     * Had New York Heart Association (NYHA) Class III-IV congestive heart failure; ③ Had a myocardial infarction or received coronary artery bypass grafting (CABG) / coronary artery stent implantation within 6 months before signing the informed consent;

       * Had clinically significant ventricular arrhythmia or a history of unexplained syncope; ⑤ Had a history of syncope (excluding cases caused by vasovagal reactions or dehydration); ⑥ Had a history of severe non-ischemic cardiomyopathy;
7. Other clinically significant diseases, including but not limited to:

   * Primary immunodeficiency; ② Had a stroke or seizure within 6 months before screening;

     * Had clear clinical evidence of dementia or mental status changes; ④ Had Parkinson's disease, Parkinson-like movement disorders or a history of the above;
8. Had undergone surgery within 2 weeks before administration, or planned to undergo surgery within 2 weeks after administration (local anesthesia surgery excluded);
9. Had received live attenuated vaccines within 1 month before administration;
10. Had a history of severe allergic reactions to this product or its formulation components;
11. Patients who were not suitable for establishing intravenous access;
12. The investigator believed that there were other conditions that made the patient unsuitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.
Incidence of adverse events(AE) after infusion | Up to 28 days after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.

SECONDARY OUTCOMES:
Objective Response Rate | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  Objective Response Rate(ORR) is defined as the proportion of subjects achieving complete remission(CR) and partial response(PR).

CONTACTS AND LOCATIONS:
Overall Officials: Wang Sanbin, MD, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No